CLINICAL TRIAL: NCT01133899
Title: The Effects of Medium-term Oral Guanidinoacetic Acid (GAA) Administration on Human Performance, Body Composition, and Metabolic Outcomes in Physically Active Men and Women
Brief Title: Guanidinoacetic Acid (GAA) Administration in Physically Active Men and Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Metropolitan University, Serbia (Other)
Responsible Party: Principal Investigator, Sergej M. OSTOJIC, Heaf of Exercise Physiology Lab, Metropolitan University, Serbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AN-85E-S09
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Athletic Performance
Keywords: strength, anaerobic performance, recovery, ergogenic
MeSH Terms: interventions — glycocyamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GAA-2 (Experimental): 2.4 grams of guanidinoacetic acid
  Interventions: Dietary Supplement: guanidinoacetic acid
- GAA-1 (Experimental): 1.2 grams of guanidinoacetic acid
  Interventions: Dietary Supplement: GAA-1
- GAA-4 (Experimental): 4.8 grams of guanidinoacetic acid
  Interventions: Dietary Supplement: GAA-4
- PLACEBO (Placebo Comparator): cellulose
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: guanidinoacetic acid — 2.4 grams of guanidinoacetic acid
  Arms: GAA-2
Dietary Supplement: GAA-4 — 4.8 grams of guanidinoacetic acid
  Arms: GAA-4
Dietary Supplement: GAA-1 — 1.2 grams of guanidinoacetic acid
  Arms: GAA-1
Dietary Supplement: PLACEBO — celulose
  Arms: PLACEBO

SUMMARY:
Glycocyamine (guanidinoacetic acid - GAA) is the biochemical precursor of creatine, which is phosphorylated and plays an important role as a high-energy carrier in the muscle. Since GAA can be administered in liquid solutions, such as sports drinks, it could be hypothesised that GAA could easily enhance creatine biosynthesis with clear physiological effects yet to be determined. No single study has examined the influence of GAA on health, human performance or body composition indicators in healthy human subjects. Moreover, the most effective dose of GAA is yet to be find. Finally, the adverse effects of GAA supplementation in humans are not determined. The main aims of the present study will be to identify if the 6-weeks of GAA supplementation improves human performance and body composition, to determine most effective dose regimens of GAA, and to analyze adverse effects of GAA supplementation. Forty eight healthy, trained (> 2 yr training experience) male and female subjects (aged 20 to 25 years) will give their informed consent and volunteer to participate in the study, which will obtain the approval of the University's Ethical Advisory Commission. The subjects will be allocated to four randomly assigned trials: ingesting GAA (1.2, 2.4, 4.8 g of GAA in a single dose) or placebo (PLA) for 6 weeks in a double-blind design. All testing including blood and urine samples, body composition and muscle strength and exercise performance (both aerobic and anaerobic) will be conducted at presupplementation (baseline), at 1 week, at 2 weeks, at 4 weeks, at 6 weeks of supplementation and at 8 and 10 weeks (2 and 4 weeks after the end of supplementation) to analyze wash-out period. According to previous investigations, the investigators expect that ingestion of GAA will significantly increase both serum creatine and total homocystein. The investigators expect that ingestion of GAA will significantly improve muscle strength parameters and exercise performance results as compared to placebo in long term. The investigators also expect to find prevalence of side-effects (i.e. gastrointestinal distress, retention of fluid).

DETAILED DESCRIPTION:
For the last two decades, top athletes first, then sport professionals and amateur sports participants have been using oral creatine supplementation on regular basis as an ergogenic aid to improve performance (Poortmans & Francaux 2000). Up to 90% of team-game athletes are regular consumers of creatine (Striegel et al. 2006), with nearly 60% of recreational athletes have tried creatine (Froiland et al. 2004). Supplementation with oral creatine, that currently is viewed to be safe, augments skeletal muscle creatine concentrations in most individuals, which has been shown to promote gains in lean body mass when used in conjunction with resistance training, to enhance power and strength, and to improve performance in intense exercise, especially during repeated bouts (Racette 2003; Ostojic 2004). Yet, creatine is not stable in solution and as such is only offered in a variety of non-liquid forms including powder, tablets, gel, chewing gum, and candy (Benzi & Ceci 2001). Although creatine synthesis is a proprietary process among manufacturers, it is quite common to use another muscle-related compounds (i.e. sarcosine, cyanamide), as the principal starting materials for the commercial synthesis of creatine (Williams & Branch 1998). Glycocyamine (guanidinoacetic acid - GAA) along with L-ornithine is formed from arginine and glycine in the kidney, with this reaction is believed to be the regulated step of creatine biosynthesis (Edison et al. 2007). The second enzyme in the pathway is GAA N-methyltransferaze which catalyzes the transfer of a methyl group from S-adenosylmethionine (SAM) to GAA to form S-adenosylhomocysteine (SAH) and creatine (Walker 1979). It has been estimated that about 75% of labile methyl groups is used to synthetize creatine by a reaction catalyzed by GAA N-methyltransferaze (Mudd et al. 1975). It seems that creatine synthesis is an interorgan process whereby GAA, produced by the kindey, is released into the circulation and is methylated to creatine in the liver. Creatine is then released from the liver and into the circulation where it can be taken up, via a specific transporter, by various tissues. According to previous studies in animals (da Silva et al. 2009) and preliminary research in humans (AlzChem 2009), short-term oral intake of GAA increases serum level of creatine, with level of increase interrelated with GAA dose supplemented. GAA is the biochemical presursor of creatine, which is phosphorylated and plays an important role as a high-energy carrier in the muscle (Edison et al. 2007). Since GAA can be administred in liquid solutions, such as sports drinks, it could be hypothesised that GAA could easily enhance creatine biosynthesis with clear physiological effects yet to be determined. Moreover, it seems that GAA has a significantly better bioavailability than creatine, developing maximal activity at a dosage at which creatine leads to no observable effects (AlzChem 2009). Several human studies (Borsook & Borsook 1951; Graybiel & Patterson 1951; Higgins et al. 1952; Dixon et al. 1954) found beneficial effects of creatine precursors oral administration on cardiac decompensation, arthritis, anxiety and depression patients. Authors speculated that benefical effects of GAA intake could be due to boosting energy levels and/or increased availability of dimethylglycine for incorporation into tissue proteins, providing repair of damaged muscle cells. Yet, no single study has examined the influence of additive-free GAA (e.g. without betaine or choline) on health, human performance or body composition indices. The amount taken of this supplementation ranges typically from a few grams to tens of grams per day for weeks or months in previous research in humans. Although, the most effective dose is yet to be find. Finally, the adverse effects of GAA supplementation in both animals and humans are yet to be determined. Several studies showed moderate hyperhomocysteinemia (Stead et al. 2001; Fukada et al. 2006; Setoue et al. 2008; AlzChem 2009), disturbances in antioxidant system (Zugno et al. 2008), modulation of inflammatory responses (Glorieux et al. 2004) after GAA supplementation. If GAA have ergogenic properties it could become new effective performance-enhancing substance for both professional and recreational athletes, stable in water solutions, where creatine at neutral to slightly acidic pH-values is rapidly being metabolised to creatinine, which is meaningless for the energy production (AlzChem 2009).

ELIGIBILITY:
Inclusion Criteria:

* healthy young men and women
* aged 20 to 25 years
* experienced in athletic training
* free from musculoskeletal dysfunctions
* free from metabolic and heart diseases
* participating in consistent training (average of three times per week)

Exclusion Criteria:

* current intake of dietary supplement containing performance-enhancing agent
* pregnant women
* current intake of hormonal contraceptives

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Muscle power | Baseline, at 1 week, at 2 weeks, at 4 weeks, at 6 weeks, at 8 weeks, at 10 weeks
  The majority of investigations involving the effects of creatine (or creatine precursors) supplementation on human performance were laboratory-based and have focused on musucular strength and power and anaerobic endurance, with various task protocols such as weght lifting, running, jumping and cycling less than or equal to 30 sec in duration. Similarly, the effects of GAA on exercise performance should be investigated with measuring muscle strength and power (through both isometric and isotonic exercise) and anaerobic endurance (e.g. repeated jumping performance).

SECONDARY OUTCOMES:
Muscle mass | Baseline, at 1 week, at 2 weeks, at 4 weeks, at 6 weeks, at 8 weeks and at 10 weeks
  A creatine supplementation-induced increase in body mass, particularly if not muscle mass, could be detrimental to performance in sports in which the body mass needs to be moved efficiently from one point to another. If GAA acts as creatine, which is an osmotically active substance, an increase in intracellular creatine concentration may likely induce influx of water into the cell. Therefore, changes of body mass and body composition (particularly muscle mass) after GAA intake should be monitored during the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Principal Investigator — Biomedical Sciences Dept, Faculty of Sport Sciences and Tourism, Metropolitan University
Locations (1):
- Biomedical Scinces Department, Exercise Physiology Lab, Novi Sad, Vojvodina, Serbia

REFERENCES:
- [Background] Setoue M, Ohuchi S, Morita T, Sugiyama K. Hyperhomocysteinemia induced by guanidinoacetic acid is effectively suppressed by choline and betaine in rats. Biosci Biotechnol Biochem. 2008 Jul;72(7):1696-703. doi: 10.1271/bbb.70791. Epub 2008 Jul 7. PMID 18603787
- [Background] Ostojic SM. Creatine supplementation in young soccer players. Int J Sport Nutr Exerc Metab. 2004 Feb;14(1):95-103. doi: 10.1123/ijsnem.14.1.95. PMID 15129933
- [Background] BORSOOK ME, BORSOOK H. Treatment of cardiac decompensation with betaine and glycocyamine. Ann West Med Surg. 1951 Oct;5(10):830-55. No abstract available. PMID 14878414
- [Background] da Silva RP, Nissim I, Brosnan ME, Brosnan JT. Creatine synthesis: hepatic metabolism of guanidinoacetate and creatine in the rat in vitro and in vivo. Am J Physiol Endocrinol Metab. 2009 Feb;296(2):E256-61. doi: 10.1152/ajpendo.90547.2008. Epub 2008 Nov 18. PMID 19017728
- [Background] Edison EE, Brosnan ME, Meyer C, Brosnan JT. Creatine synthesis: production of guanidinoacetate by the rat and human kidney in vivo. Am J Physiol Renal Physiol. 2007 Dec;293(6):F1799-804. doi: 10.1152/ajprenal.00356.2007. Epub 2007 Oct 10. PMID 17928413
- [Background] Mudd SH, Poole JR. Labile methyl balances for normal humans on various dietary regimens. Metabolism. 1975 Jun;24(6):721-35. doi: 10.1016/0026-0495(75)90040-2. PMID 1128236
- [Derived] Ostojic SM, Stojanovic M, Drid P, Hoffman JR. Dose-response effects of oral guanidinoacetic acid on serum creatine, homocysteine and B vitamins levels. Eur J Nutr. 2014 Dec;53(8):1637-43. doi: 10.1007/s00394-014-0669-0. Epub 2014 Feb 18. PMID 24535415
- [Derived] Ostojic SM, Niess B, Stojanovic M, Obrenovic M. Creatine metabolism and safety profiles after six-week oral guanidinoacetic acid administration in healthy humans. Int J Med Sci. 2013;10(2):141-7. doi: 10.7150/ijms.5125. Epub 2013 Jan 3. PMID 23329885